CLINICAL TRIAL: NCT00182975
Title: Is DHEA Replacement Beneficial?
Brief Title: Effects of Dehydroepiandrosterone (DHEA) in Humans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG0047; R01AG020076 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Aging
Keywords: Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

INTERVENTIONS:
Drug: DHEA replacement

SUMMARY:
The purpose of this study is to determine whether bringing back the DHEA levels of older persons to the young range produces beneficial effects.

DETAILED DESCRIPTION:
DHEA and DHEA sulfate (DHEAS) plasma concentrations peak at about 20 years of age and decline rapidly and markedly after age 25 yr. DHEA is a PPAR-alpha activator. PPAR-alpha plays major roles in regulating lipid metabolism and controlling inflammation. DHEA also appears to have anabolic effects on muscle and bone. The study is designed to determine the effects of 12 months of DHEA replacement in 65-75 year old women and men on (a) truncal and visceral fat, (b) insulin resistance and serum triglycerides, (c) muscle mass and strength, (d) bone mineral density, (e) chronic inflammation, (f) arterial-endothelium-dependent vasodilation, and (g) sense of well being.

The specific aims of this study are to test the hypotheses that 12 months of DHEA replacement will (a) Result in significant decreases in truncal and visceral fat by shifting metabolism to fat oxidation and increasing energy wastage; (b) Decrease insulin resistance and decrease serum triglycerides; (c) Increase muscle mass and strength, by decreasing catabolic stimuli and increasing anabolic stimuli; (d) Increase bone mineral density by increasing anabolic stimuli and decreasing catabolic stimuli; (e) Reduce chronic inflammation and decrease pro-inflammatory cytokine production by peripheral blood mononuclear cells; (f) Improve arterial endothelium dependent vasodilation; and (g) Improve general sense of well being.

ELIGIBILITY:
Inclusion Criteria:

* 65 to 75 years old
* Physically healthy
* Non-smoker
* On stable medications for at least 6 months
* Stable body weight for the past year

Exclusion Criteria:

* Serious active medical problems
* Hormone therapy
* Abnormal PSA (prostate specific antigen) in men

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 142 (Actual)
Dates: Start 2002-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
body composition (e.g. truncal fat and visceral fat), insulin resistance and serum triglycerides, muscle mass and strength

SECONDARY OUTCOMES:
bone mineral density, arterial-endothelium dependent vasodilatation, sense of well being, RMR (Resting Metabolic Rate), TEF (Thermal Effect of Food)

CONTACTS AND LOCATIONS:
Overall Officials: John O. Holloszy, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Hansen PA, Han DH, Nolte LA, Chen M, Holloszy JO. DHEA protects against visceral obesity and muscle insulin resistance in rats fed a high-fat diet. Am J Physiol. 1997 Nov;273(5):R1704-8. doi: 10.1152/ajpregu.1997.273.5.R1704. PMID 9374813
- [Background] Han DH, Hansen PA, Chen MM, Holloszy JO. DHEA treatment reduces fat accumulation and protects against insulin resistance in male rats. J Gerontol A Biol Sci Med Sci. 1998 Jan;53(1):B19-24. doi: 10.1093/gerona/53a.1.b19. PMID 9467418
- [Background] Villareal DT, Holloszy JO, Kohrt WM. Effects of DHEA replacement on bone mineral density and body composition in elderly women and men. Clin Endocrinol (Oxf). 2000 Nov;53(5):561-8. doi: 10.1046/j.1365-2265.2000.01131.x. PMID 11106916
- [Derived] Weiss EP, Shah K, Fontana L, Lambert CP, Holloszy JO, Villareal DT. Dehydroepiandrosterone replacement therapy in older adults: 1- and 2-y effects on bone. Am J Clin Nutr. 2009 May;89(5):1459-67. doi: 10.3945/ajcn.2008.27265. Epub 2009 Mar 25. PMID 19321570